CLINICAL TRIAL: NCT05319548
Title: Plant Pigments for Human Health: Determining the Interactions the Impact of Co-ingestion of Carotenoids and Anthocyanins From Multicolored Carrots on the Bioavailability of Provitamin A Carotenoids and the Impact on Each Pigment Groups' Respective Antidiabetic Activity in Humans
Brief Title: Plant Pigments for Human Health: Impact of Lycopene and Anthocyanins on Bioefficacy of Provitamin A Carotenoids From Carrots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-1544; Protocol Version 6/9/2022 (Other: UW Madison); A074600 (Other: UW Madison); 59-5090-2-003 (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2022-03-29; First posted 2022-04-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Starting with Purple-Red Carrot Juice (Active Comparator): Participants are randomized to consume purple-red carrot juice first (250 mL) in under 2 minutes. They will crossover to red carrot juice and to purple carrot juice.
  Interventions: Other: Purple-Red Carrot Juice; Other: Red Carrot Juice; Other: Purple Carrot Juice
- Starting with Purple Carrot Juice (Active Comparator): Participants are randomized to consume purple carrot juice first (250 mL) in under 2 minutes. They will crossover to red carrot juice and to purple-red carrot juice.
  Interventions: Other: Purple-Red Carrot Juice; Other: Red Carrot Juice; Other: Purple Carrot Juice
- Starting with Red Carrot Juice (Active Comparator): Participants are randomized to consume red carrot juice first (250 mL) in under 2 minutes. They will crossover to purple-red carrot juice and to purple carrot juice.
  Interventions: Other: Purple-Red Carrot Juice; Other: Red Carrot Juice; Other: Purple Carrot Juice

INTERVENTIONS:
Other: Purple-Red Carrot Juice — Purple-Red carrot juice contains provitamin A carotenoids (beta-carotene, alpha-carotene), the non-provitamin A carotenoid, lycopene, as well as anthocyanins
Other: Red Carrot Juice — Red carrot juice contains provitamin A carotenoids (beta-carotene, alpha-carotene), and the non-provitamin A carotenoid, lycopene, but does NOT contain anthocyanins..
Other: Purple Carrot Juice — Purple carrot juice does NOT contain provitamin A carotenoids (beta-carotene, alpha-carotene), nor the non-provitamin A carotenoid, lycopene, but contains anthocyanins.

SUMMARY:
The proposed research will help characterize the impact that simultaneous consumption of anthocyanins and carotenoids has on the bioavailability of the provitamin A carotenoids a-carotene and b-carotene and the non-provitamin A carotenoid lycopene, and on their respective antidiabetic activity in humans. The central hypothesis is that provitamin A carotenoids will be bioavailable from purple-red multicolored carrots in humans, and the co-ingestion of carotenoids and anthocyanins from these carrots will have synergistic impacts on their respective antioxidant and antidiabetic effects. This hypothesis will be assessed through a 53 day randomized crossover time course study that consists of three arms in which healthy males and females ages 18-40 (n = 12) will consume carrot juice prepared from red, purple-red, or purple carrots. During each arm, participants will switch the type of juice they consume and by the end of the third arm, all participants will have ingested juice made from all three carrot varieties. Blood will be collected at multiple time points over 72 hours following consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking
* Not pregnant (or planning to become pregnant)
* Body Mass Index (BMI) greater than 18.5 and less than 30

Exclusion Criteria:

* Major comorbidities (cardiovascular disease (CVD), diabetes, cancer, kidney/liver/bowel disease)
* History of malabsorptive/GI disorders
* Abnormal diet
* BMI less than 18.5 or greater than 30
* Food intolerances/allergies/hypersensitivities
* History of substance abuse or alcoholism
* Unwilling to restrict consumption of specific foods prior to study
* Unwilling to participate in blood draws
* History of difficulty drawing blood/health issues associated with blood draws (gets dizzy, etc).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Change in serum retinol concentration | Blood will be drawn on the first test day (treatment day) at baseline, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2.5 hours, 4 hours, 6 hours, 9 hours, 24 hours, 72 hours
  Blood draws will take place on the first, second, and fourth test day (days 8, 9, 11 of each arm)
Change in serum carotenoid concentration | Blood will be drawn on the first test day (treatment day) at baseline, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2.5 hours, 4 hours, 6 hours, 9 hours, 24 hours, 72 hours
  Blood draws will take place on the first, second, and fourth test day (days 8, 9, 11 of each arm)
Change in serum anthocyanin concentration | Blood will be drawn on the first test day (treatment day) at baseline, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2.5 hours, 4 hours, 6 hours, 9 hours, 24 hours, 72 hours
  Blood draws will take place on the first, second, and fourth test day (days 8, 9, 11 of each arm)

SECONDARY OUTCOMES:
Change in antioxidant capacity of the carrots and carrot juice measured by enzyme activity assay | up to 1 month
  Three different antioxidant activity assays will be used including the Oxygen Radical Absorbance Capacity (ORAC), 2,2'-azino-bis-3-ethylbenzthiazoline-6-sulphonic acid (ABTS+), and 1,1-diphenyl-2-picrylhydrazyl (DPPH) assays, all of which will be analyzed by Ultraviolet (UV) spec. Each method analyzes different ways anthocyanins and carotenoids may act as antioxidants, and a combination of the three will more accurately represent the parameters of human biology. Data will be expressed as Trolox equivalent antioxidant capacity (TEAC).
Change in alpha-glucosidase inhibition activities of the carrots and carrot juice measured by enzyme activity assay | up to 1 month
  Enzyme inhibition will be assessed using specific enzymatic assay kits for alpha-glucosidase and alpha-amylase, analyzed using Enzyme-Linked Immunosorbent Assay (ELISA), and results will be expressed as IC50 (% inhibition).
Change in alpha-amylase inhibition activities of the carrots and carrot juice measured by enzyme activity assay | up to 1 month
  Enzyme inhibition will be assessed using specific enzymatic assay kits for alpha-glucosidase and alpha-amylase, analyzed using ELISA, and results will be expressed as IC50 (% inhibition).
Change in serum glucose concentration | Blood will be drawn on the first test day (treatment day) at baseline, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2.5 hours, 4 hours, 6 hours, 9 hours, 24 hours, 72 hours
  Blood draws will take place on the first, second, and fourth test day (days 8, 9, 11 of each arm)
Change in serum insulin concentration | Blood will be drawn on the first test day (treatment day) at baseline, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2.5 hours, 4 hours, 6 hours, 9 hours, 24 hours, 72 hours
  Blood draws will take place on the first, second, and fourth test day (days 8, 9, 11 of each arm)
Change in serum incretin concentration | Blood will be drawn on the first test day (treatment day) at baseline, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2.5 hours, 4 hours, 6 hours, 9 hours, 24 hours, 72 hours
  Blood draws will take place on the first, second, and fourth test day (days 8, 9, 11 of each arm)

CONTACTS AND LOCATIONS:
Locations (1):
- UW-Madison Department of Nutritional Sciences, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT05319548/ICF_000.pdf